CLINICAL TRIAL: NCT04819152
Title: Effectiveness of Tobacco Cessation Interventions for Different Groups of Users in Sweden: a National Prospective Cohort Study
Brief Title: Effectiveness of Tobacco Cessation Interventions in Sweden
Acronym: RSP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Hanne Tonnesen, Professor, Lund University
Other Study IDs: Rökstoppsprojektet; Dnr: 2019-02221 (Other: Etikprövningsmyndigheten); 2017-01681 (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Tobacco Use; Smoking; Cigarette Use, Electronic
Keywords: National cohort study; Effectiveness; Tobacco use cessation; Smoking cessation; Vulnerable groups
MeSH Terms: conditions — Tobacco Use; Smoking; Vaping; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Several studies will be performed based on this cohort. I each study the exposed group will be a group of tobacco users evaluatedin the relevant study. This could be a vulnarable group tobacco users such as: users without a job, with short or no education, without permanent housing, diagnosed with mental illness, diagnosed with chronic obstructive pulmonary disease (COPD), undergoing surgery, adolescents, elderly, migrants, or pregnant women.
  Interventions: Behavioral: Tobacco cessation intervention
- Unexposed: In each study the unexposed group will consist of tobacco user from the study cohort without the condition examined in the relevant study.
  Interventions: Behavioral: Tobacco cessation intervention

INTERVENTIONS:
Behavioral: Tobacco cessation intervention — Already implemented in-person (including online meetings) tobacco cessation interventions in Sweden

SUMMARY:
Smoking is still one of the most important risk factors causing morbidity and mortality in Sweden. Every year, 12,000 Swedish citizens die prematurely from smoking, and smoking is responsible for up to 60% of the inequity in health.

Though the smoking prevalence is relatively low in Sweden in an international context (8% and 10% for men and women respectively in 2016), specific vulnarable groups have a very high prevalence; e.g. about 80% in alcohol and drug abusers. Furthermore, Sweden has a unique high prevalence of snus users and in 2016 the daily use of tobacco was 25% for men and 14% for women. In addition, products such as cigarettes, snus, and e-cigettes are often mixed.

Despite the fact that about a thousand counsellors have been trained in manual-based person-centred tobacco cessation interventions in Sweden, the effectiveness of the interventions remains unknown, as a follow-up on effect of in-person interventions is not systematically collected in Sweden. Therefore, as of today it is not possible, on a national level, to compare the effectiveness of differences in these interventions, providers, or different groups of tobacco users including disadvantaged and vulnerable groups.

In this study the investigators will evaluate the effectiveness of already implemented in-person cessation interventions targeting smoking, use of snus and/or e-cigarettes, focusing on disadvantaged and vulnerable groups of tobacco users. Furthermore, important factors associated with a successful outcome after controlling for confounders will be identified (in relation to programme, patients and setting).

ELIGIBILITY:
Inclusion Criteria:

* All adult tobacco users (of at least 18 years of age), including disadvantaged and vulnerable patients, receiving an in-person intervention (incl. online meetings) for tobacco cessation (smoking, snus and/or e-cigarettes) are eligible for inclusion in the project after giving informed consent.
* Both individual and group-based interventions can be included.

Exclusion Criteria:

* Withdrawing consent.
* Reduced ability to give informed consent, due to inadequate language skills, dementia, and other conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population in this study are tobacco users in Sweden, who have attented an in-person tobacco cessation programme.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
% of patients that are continuously smokefree | 6 months
  Self-reported smoking status, questionnaire completed by telephone interview

SECONDARY OUTCOMES:
% of patients that are smokefree | On completion of the tobacco cessation programme (app. 1 month after quitting)
  Counsellor observed smoking status, questionnaire completed by counsellor
% of patients that have been smokefree for at least the latest 14 days | 6 months
  Self-reported smoking status, questionnaire completed by telephone interview
% of patients that are satisfied with the smoking cessation intervention | 6 months
  Self-reported patient-satisfaction, questionnaire completed by telephone interview

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Tønnesen, DSc, Principal Investigator — Lund University, Clinical health promotion centre
Locations (8):
- Sweden (8):
  - Tobaksavvänjningen, Kirurgisk mott., CLV Växjö lasarett, Vaxjo, Kronoberg County
  - Capio Go, Malmo, Skåne County
  - Livsstilsmedicin Österåsen, Sollefteå, Västernorrland County
  - Tobakspreventiva enheten, USÖ, Örebro
  - Tybble vårdcentral, Örebro
  - Ekeby Hälsocenter, Uppsala
  - Flogsta vårdcentral, Uppsala
  - Tobakspreventiv mottagning Karlskoga, Karlskoga, Örebro County

REFERENCES:
- [Background] Rasmussen M, Larsson M, Gilljam H, Adami J, Warjerstam S, Post A, Bjork-Eriksson T, Helgason AR, Tonnesen H. Effectiveness of tobacco cessation interventions for different groups of tobacco users in Sweden: a study protocol for a national prospective cohort study. BMJ Open. 2022 Jan 25;12(1):e053090. doi: 10.1136/bmjopen-2021-053090. PMID 35078840